CLINICAL TRIAL: NCT04497389
Title: A Phase I/II Randomized Double-blinded Placebo-controlled Clinical Trial to Determine Safety and Feasibility of Using an Acellular Sterile Filtered Amniotic Fluid as a Treatment for COVID-19 Patients
Brief Title: Safety and Feasibility of Amniotic Fluid as a Treatment for COVID-19 Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Craig Selzman, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 132922
Record Dates: First submitted 2020-06-09; First posted 2020-08-04 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: SARS CoV-2
Keywords: Amniotic fluid; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — amniotic fluid peptide-1, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): 10ml intravenous hAF QD (once daily) for 5 consecutive days
  Interventions: Biological: Human Amniotic Fluid
- Standard of Care (No Intervention): 10 mL normal saline QD (once daily) for 5 days

INTERVENTIONS:
Biological: Human Amniotic Fluid — Patients will receive 10ml intravenous hAF each day for 5 consecutive days.
  Arms: Intervention

SUMMARY:
The purpose of this study is to explore the effectiveness of processed human amniotic fluid as a treatment for COVID-19.

DETAILED DESCRIPTION:
Past use of human amniotic products (i.e., membrane and fluid) has previously been FDA-approved as a human cells, Tissues, and Cellular and Tissue-Based Products (HCT/P) under 21 CFR 1271 for tissue injury; and has been used to reduce inflammation and fibrosis in patients with a variety of ailments. Given this, the investigators hypothesize that intravenously (IV) administered processed sterile filtered amniotic fluid will reduce inflammation in COVID-19 patients, and improve secondary clinical outcomes. Specifically, the investigators hypothesize that patients who receive IV administered hAF will see a 50% reduction in mean C-reactive protein levels following treatment.

Data sharing: Trial results will be published in peer reviewed publications upon completion of analysis.

ELIGIBILITY:
Inclusion criteria:

1. Age >18
2. SARS CoV-2 laboratory positive test, obtained within 14 days of enrollment
3. Hospitalized
4. COVID-19 symptomatic (cough, fevers, shortness of breath, and/or sputum production)
5. Has a room air pulse oximetry of ≤94% and requires supplemental oxygen therapy
6. Patients of childbearing potential who agree to use acceptable methods of contraception for 90 days after last administration of study investigational product (IP)
7. Patients who are receiving standard of care therapies for COVID-19 that are not FDA approved are eligible for this study
8. Subjects must be able to consent to the study (i.e., Glasgow Coma Scale score of ≥14)
9. Patients are required to have controlled blood pressure of <160/96 and a pulse of <110.

Exclusion criteria:

1. Patients on invasive mechanical ventilation (e.g., endotracheal intubation)
2. Chronic home oxygen utilization
3. Home or current use of immunosuppressive medications (including steroids)
4. Women who are pregnant, breastfeeding, or become pregnant during the study
5. Patients on non-invasive positive pressure ventilation
6. Patients on >12 liters per minute via non-rebreather (NRB) or >80% oxygen via high flow nasal cannula
7. Patients who, in the opinion of the PI, have impending respiratory failure, defined as requiring rapidly escalating oxygen supplementation
8. Patients with a hemoglobin <9 mg/dL
9. Patients diagnosed with Stage 4 or 5 chronic kidney disease (CKD)
10. Patients with diagnosed New York Heart Association (NYHA) class 4 or 5 congestive heart failure
11. Patients with a left ventricular assist device (LVAD)
12. Patients with thromboembolic phenomena
13. Patients with Type 2 and above heart block
14. Patients with established positive bacterial blood cultures prior to enrollment
15. Patients with ongoing pericardial effusion or ascites
16. Patients with clinically significant arrhythmia
17. Patients with liver function tests (ALT or AST) >3x normal
18. Patients with untreated HIV infection
19. Patients diagnosed with end-stage organ disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Selzman, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Tonna JE, Pierce J, Brintz BJ, Bardsley T, Hatton N, Lewis G, Phillips JD, Skidmore CR, Selzman CH. A randomized, double-blinded, placebo-controlled clinical trial of sterile filtered human amniotic fluid for treatment of COVID-19. BMC Infect Dis. 2023 Dec 8;23(1):864. doi: 10.1186/s12879-023-08856-y. PMID 38066442
- [Derived] Tonna JE, Pierce J, Hatton N, Lewis G, Phillips JD, Messina A, Skidmore CR, Taylor K, Selzman CH. Safety and feasibility of using acellular sterile filtered amniotic fluid as a treatment for patients with COVID-19: protocol for a randomised, double-blinded, placebo-controlled clinical trial. BMJ Open. 2021 Feb 11;11(2):e045162. doi: 10.1136/bmjopen-2020-045162. PMID 33574155

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: 10ml intravenous hAF QD for 5 consecutive days
  Human Amniotic Fluid: Patients will receive 10ml intravenous hAF each day for 5 consecutive days.
- Standard of Care: 10 mL normal saline QD for 5 days
Period: Overall Study
Arm/Group | Intervention | Standard of Care
Started | 23 | 24
Completed | 22 | 24
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard of Care | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (16.09) | 58.8 (12.8) | 57.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 0 | 1 | 1
  White | 15 | 19 | 34
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: C-reactive Protein
Description: Assess reduction of inflammation in COVID-19 patients, potentially leading to a decrease in the need for critical care. This will be assessed by measurement of C-reactive protein levels before and after the intervention. Units: mg/dL
Time Frame: Baseline through post-treatment (6 days)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 23 | 24
mg/dL | -3.6 (8.58) | -5.5 (5.42)

2. Other Pre Specified Outcome: Death Within 30 Days
Description: Comparison of mortality between intervention and control groups
Time Frame: Baseline through 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 23 | 24
Participants | 2 | 0

3. Other Pre Specified Outcome: Any ICU Admission
Description: Comparison of ICU admissions between intervention and control groups
Time Frame: Baseline through 30 days
Measure: Number; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 22 | 24
Participants | 8 | 4

4. Other Pre Specified Outcome: Hospital Length of Stay
Description: Comparison of days spent in hospital between intervention and control groups
Time Frame: From date of hospital admission through date of discharge or death, whichever comes first (up to 100 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 23 | 24
days | 7.4 (6.69) | 7 (6.04)

5. Other Pre Specified Outcome: Need for Invasive Mechanical Ventilation
Description: Comparison of mechanical ventilation incidence between intervention and control groups
Time Frame: From date of enrollment through date of discharge or death, whichever comes first (up to 100 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 23 | 24
Participants | 4 | 1

6. Other Pre Specified Outcome: Biomarker Levels (Interleukin-6)
Description: Comparison of mean biomarker level change between intervention and control groups. Units: pg/mL
Time Frame: Baseline through post-treatment (6 days)
Population: Data is missing for patients who did not have Day 6 labs drawn.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 17 | 15
pg/mL | 9.4 (24.11) | 32 (107.77)

7. Other Pre Specified Outcome: Biomarker Levels (D-dimer)
Description: Comparison of mean biomarker level change between intervention and control groups. Units: mg/mL
Time Frame: Baseline through post-treatment (6 days)
Population: Data is missing for patients who did not have Day 6 labs drawn.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 19 | 16
mg/mL | -0.3 (1.77) | 1.8 (11.8)

8. Other Pre Specified Outcome: Biomarker Levels (Lactate Dehydrogenase)
Description: Comparison of mean biomarker level change between intervention and control groups. Units: u/L
Time Frame: Baseline through post-treatment (6 days)
Population: Data is missing for patients who did not have Day 6 labs drawn.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 18 | 14
U/L | -87.3 (124.8) | -54.4 (80.8)

9. Other Pre Specified Outcome: Need for ECMO
Description: Comparison of ECMO incidence between intervention and control groups
Time Frame: From date of enrollment through date of discharge or death, whichever comes first (up to 100 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 23 | 24
Participants | 0 | 0

10. Other Pre Specified Outcome: Major Adverse Cardiac Events
Description: Compare frequency of major adverse cardiac events (MACE) between intervention and control groups
Time Frame: From date of enrollment through date of discharge or death, whichever comes first (up to 100 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 23 | 24
Participants | 1 | 0

11. Other Pre Specified Outcome: Patient-reported Functional Status at 1 Month
Description: Comparison of PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire results on a computer-adaptive platform between intervention and control groups using T-scores. Scale mean = 50, standard deviation = 10. Higher scores indicate more of the concept being measured (i.e., physical function = a higher score indicates better outcomes; dyspnea severity, sleep disturbance, anxiety = a higher score indicates worse outcomes).
  Sleep Disturbance, Dyspnea Severity, Anxiety Less than 55 = None to slight/Within normal limits 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe
  Physical Function 55 and over = Within normal limits 54.9-40 = Mild limitations 39.9-30 = Moderate limitations 29.9 and below = Severe limitations
Time Frame: 1 month post-discharge
Population: Data is missing for patients who did not complete Month 1 surveys.
Measure: Mean (Standard Deviation); unit: t-score
Groups:
- Month 1 PROMIS Physical Function: Intervention; Month 1 PROMIS Dyspnea Severity: Control: Results from self-reported PROMIS Physical Function at 1 month post-discharge, intervention group
- Month 1 PROMIS Physical Function: Control: Results from self-reported PROMIS Physical Function at 1 month post-discharge, control group
- Month 1 PROMIS Dyspnea Severity: Intervention: Results from self-reported PROMIS Dyspnea Severity at 1 month post-discharge, intervention group
- Month 1 PROMIS Sleep Disturbance: Intervention: Results from self-reported PROMIS Sleep Disturbance at 1 month post-discharge, intervention group
- Month 1 PROMIS Sleep Disturbance: Control: Results from self-reported PROMIS Sleep Disturbance at 1 month post-discharge, control group
- Month 1 PROMIS Anxiety: Intervention: Results from self-reported PROMIS Anxiety at 1 month post-discharge, intervention group
- Month 1 PROMIS Anxiety: Control: Results from self-reported PROMIS Anxiety at 1 month post-discharge, control group
Arm/Group | Month 1 PROMIS Physical Function: Intervention | Month 1 PROMIS Physical Function: Control | Month 1 PROMIS Dyspnea Severity: Intervention | Month 1 PROMIS Dyspnea Severity: Control | Month 1 PROMIS Sleep Disturbance: Intervention | Month 1 PROMIS Sleep Disturbance: Control | Month 1 PROMIS Anxiety: Intervention | Month 1 PROMIS Anxiety: Control
Number analyzed (Participants) | 11 | 13 | 11 | 13 | 11 | 13 | 11 | 13
t-score | 39.8 (8.54) | 41.5 (9.10) | 41.6 (9.36) | 43.0 (9.71) | 47.8 (9.81) | 52.2 (4.98) | 47.0 (9.18) | 51.1 (47.0)

12. Other Pre Specified Outcome: Patient-reported Functional Status at 3 Months
Description: as for outcome 11
Time Frame: 3 months post-discharge
Population: Data is missing for patients who did not complete Month 3 surveys.
Measure: Mean (Standard Deviation); unit: t-score
Groups:
- Month 3 PROMIS Physical Function: Intervention: Results from self-reported PROMIS Physical Function at 3 month post-discharge: intervention group
- Month 3 PROMIS Physical Function: Control: Results from self-reported PROMIS Physical Function at 3 month post-discharge: control group
- Month 3 PROMIS Dyspnea Severity: Intervention: Results from self-reported PROMIS Dyspnea Severity at 3 month post-discharge: intervention group
- Month 3 PROMIS Dyspnea Severity: Control: Results from self-reported PROMIS Dyspnea Severity at 3 month post-discharge: control group
- Month 3 PROMIS Sleep Disturbance: Intervention: Results from self-reported PROMIS Sleep Disturbance at 3 month post-discharge: intervention group
- Month 3 PROMIS Sleep Disturbance: Control: Results from self-reported PROMIS Sleep Disturbance at 3 month post-discharge: Control group
- Month 3 PROMIS Anxiety: Intervention: Results from self-reported PROMIS Anxiety at 3 month post-discharge: intervention group
- Month 3 PROMIS Anxiety: Control: Results from self-reported PROMIS Anxiety at 3 month post-discharge: control group
Arm/Group | Month 3 PROMIS Physical Function: Intervention | Month 3 PROMIS Physical Function: Control | Month 3 PROMIS Dyspnea Severity: Intervention | Month 3 PROMIS Dyspnea Severity: Control | Month 3 PROMIS Sleep Disturbance: Intervention | Month 3 PROMIS Sleep Disturbance: Control | Month 3 PROMIS Anxiety: Intervention | Month 3 PROMIS Anxiety: Control
Number analyzed (Participants) | 11 | 13 | 11 | 13 | 11 | 13 | 11 | 13
t-score | 42.9 (7.30) | 43.9 (10.4) | 37.2 (10.3) | 41.5 (14.8) | 45.4 (10.8) | 50.5 (8.55) | 43.6 (6.87) | 50.9 (7.84)

13. Other Pre Specified Outcome: Patient-reported Functional Status at 6 Months
Description: as for outcome 11
Time Frame: 6 months post-discharge
Population: Data is missing for patients who did not complete Month 6 surveys.
Measure: Mean (Standard Deviation); unit: t-score
Groups:
- Month 6 PROMIS Physical Function: Intervention: Results from self-reported PROMIS Physical Function at 6 month post-discharge: Intervention group
- Month 6 PROMIS Physical Function: Control: Results from self-reported PROMIS Physical Function at 6 month post-discharge: Control group
- Month 6 PROMIS Dyspnea Severity: Intervention: Results from self-reported PROMIS Dyspnea Severity at 6 month post-discharge: Intervention group
- Month 6 PROMIS Dyspnea Severity: Control: Results from self-reported PROMIS Dyspnea Severity at 6 month post-discharge: Control group
- Month 6 PROMIS Sleep Disturbance: Intervention: Results from self-reported PROMIS Sleep Disturbance at 6 month post-discharge: Intervention group
- Month 6 PROMIS Sleep Disturbance: Control: Results from self-reported PROMIS Sleep Disturbance at 6 month post-discharge: Control group
- Month 6 PROMIS Anxiety: Intervention: Results from self-reported PROMIS Anxiety at 6 month post-discharge: Intervention group
- Month 6 PROMIS Anxiety: Control: Results from self-reported PROMIS Anxiety at 6 month post-discharge: Control group
Arm/Group | Month 6 PROMIS Physical Function: Intervention | Month 6 PROMIS Physical Function: Control | Month 6 PROMIS Dyspnea Severity: Intervention | Month 6 PROMIS Dyspnea Severity: Control | Month 6 PROMIS Sleep Disturbance: Intervention | Month 6 PROMIS Sleep Disturbance: Control | Month 6 PROMIS Anxiety: Intervention | Month 6 PROMIS Anxiety: Control
Number analyzed (Participants) | 8 | 11 | 8 | 11 | 8 | 11 | 8 | 11
t-score | 45.0 (6.30) | 44.3 (11.6) | 37.6 (9.21) | 37.2 (10.8) | 48.0 (10.2) | 47.1 (6.84) | 39.4 (3.23) | 51.7 (8.46)

14. Other Pre Specified Outcome: Patient-reported Functional Status at 12 Months
Description: as for outcome 11
Time Frame: 12 months post-discharge
Population: Data missing from patients who did not complete Month 12 surveys.
Measure: Mean (Standard Deviation); unit: t-score
Groups:
- Month 12 PROMIS Physical Function: Intervention: Results from self-reported PROMIS Physical Function at 12 months: Intervention group
- Month 12 PROMIS Physical Function: Control: Results from self-reported PROMIS Physical Function at 12 months: Control group
- Month 12 PROMIS Dyspnea Severity: Intervention: Results from self-reported PROMIS Dyspnea Severity at 12 months: Intervention group
- Month 12 PROMIS Dyspnea Severity: Control: Results from self-reported PROMIS Dyspnea Severity at 12 months: Control group
- Month 12 PROMIS Sleep Disturbance: Intervention: Results from self-reported PROMIS Sleep Disturbance at 12 months: Intervention group
- Month 12 PROMIS Sleep Disturbance: Control: Results from self-reported PROMIS Sleep Disturbance at 12 months: Control group
- Month 12 PROMIS Anxiety: Intervention: Results from self-reported PROMIS Anxiety at 12 months: Intervention group
- Month 12 PROMIS Anxiety: Control: Results from self-reported PROMIS Anxiety at 12 months: Control group
Arm/Group | Month 12 PROMIS Physical Function: Intervention | Month 12 PROMIS Physical Function: Control | Month 12 PROMIS Dyspnea Severity: Intervention | Month 12 PROMIS Dyspnea Severity: Control | Month 12 PROMIS Sleep Disturbance: Intervention | Month 12 PROMIS Sleep Disturbance: Control | Month 12 PROMIS Anxiety: Intervention | Month 12 PROMIS Anxiety: Control
Number analyzed (Participants) | 5 | 11 | 5 | 11 | 5 | 11 | 5 | 11
t-score | 51.8 (9.66) | 42.9 (10.9) | 31.8 (8.62) | 41.6 (12.3) | 47.1 (12.6) | 49.9 (7.64) | 42.3 (5.73) | 47.4 (9.38)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 5/23 | 2/24
Other Adverse Events (participants affected / at risk) | 13/23 | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=23) | Standard of Care (N=24)
Shock leading to death (General disorders) | 1 (1) | 0 (0) — Multifactorial shock requiring use of multiple vasopressors. Resulted in patient's death.
Shock leading to readmission (General disorders) | 1 (1) | 0 (0) — Septic shock leading to patient's readmission to the hospital.
STEMI (Cardiac disorders) | 1 (1) | 0 (0) — STEMI which resulted in patient's death
Readmission for COVID-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Continued symptoms of COVID-19 pneumonia requiring hospital readmission
Readmission for ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient developed acute respiratory distress syndrome (ARDS) which required readmission to hospital
Readmission for COVID-19 symptoms (General disorders) | 0 (0) | 1 (1) — Patient was experiencing continued COVID-19 symptoms and was readmitted to the hospital.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=23) | Standard of Care (N=24)
Abnormal Metabolic Panel (Metabolism and nutrition disorders) | 4 (9) | 2 (4) — High or low values in basic or comprehensive metabolic panels
Abnormal CBC (Blood and lymphatic system disorders) | 4 (5) | 3 (4) — Low or high values in complete blood count panel
Abnormal Hepatic Panel (Hepatobiliary disorders) | 1 (7) | 2 (4) — Low or high values on hepatic blood panel
Elevated Blood Pressure (Cardiac disorders) | 1 (2) | 0 (0) — Elevated systolic and/or diastolic blood pressure values
Hypotension (Cardiac disorders) | 5 (27) | 4 (7) — Low systolic and/or diastolic blood pressure values
Tachycardia (Cardiac disorders) | 5 (9) | 3 (6) — Heart rates above 100 beats per minute
Bradycardia (Cardiac disorders) | 3 (4) | 4 (8) — Heart rate less than 60 beats per minute
ED visits (General disorders) | 2 (3) | 1 (1) — Visits to the Emergency Department that did not result in hospital admission (e.g., ongoing cough)
Positive urine culture (Renal and urinary disorders) | 2 (2) | 0 (0) — Bacteria found in urine culture
Abnormal Blood Gas (General disorders) | 2 (30) | 1 (2) — Low or high arterial or venous blood gas values
Intubation (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) — Patients requiring endotracheal intubation
Elevated troponin (Cardiac disorders) | 2 (2) | 0 (0) — Elevated blood troponin values
Abnormal ECG (Cardiac disorders) | 1 (1) | 0 (0) — Abnormal results on electrocardiogram (e.g., bundle branch block)
Abnormal Echocardiogram (Cardiac disorders) | 2 (2) | 0 (0) — Abnormal results on echocardiogram (e.g., Takotsubo cardiomyopathy)
Fall (General disorders) | 1 (1) | 0 (0) — Patient fell while inpatient
Type 2 Diabetes (Endocrine disorders) | 1 (1) | 0 (0) — New diagnosis of Type 2 diabetes
Positive respiratory cultures (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Bacterial findings in respiratory culture
Back pain (General disorders) | 1 (1) | 0 (0) — Patient complaint of back pain while inpatient
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — Development of pneumothorax
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient complaint of abdominal pain while inpatient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04497389/Prot_SAP_000.pdf